CLINICAL TRIAL: NCT05195944
Title: The GLP-1 Agonist Semaglutide for the Treatment of Metabolic Disease in Liver Transplant Recipients: A Phase IV, Randomized Trial
Brief Title: Semaglutide vs Sitagliptin
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University Health Network, Toronto (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21-5640; U1111-1268-1934 (Registry Identifier: WHO UTN)
Record Dates: First submitted 2021-12-13; First posted 2022-01-19 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Liver Transplant; Complications; Diabetes Mellitus; NASH - Nonalcoholic Steatohepatitis; NAFLD
MeSH Terms: conditions — Diabetes Mellitus; Non-alcoholic Fatty Liver Disease | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Semaglutide (Experimental): In the Semaglutide Arm, participants will receive daily: 1 tablet of Semaglutide and 1 tablet of Sitagliptin placebo for 26 weeks. The dosages of Semaglutide are 3 mg, 7 mg, and 14 mg.
  Interventions: Drug: Semaglutide Treatment
- Sitagliptin (Active Comparator): In the Sitagliptin arm, participants will receive daily: 1 tablet of 100 mg Sitagliptin and 1 tablet of Semaglutide placebo for 26 weeks.
  Interventions: Drug: Sitagliptin 100mg

INTERVENTIONS:
Drug: Semaglutide Treatment — The participants will be provided with Semaglutide, titrated up to 14 mg. The starting dose of Semaglutide is 3 mg once daily. At week 4, the dose will be increased to 7 mg once daily. At week 8, the dose will be increased to 14 mg once daily and will be maintained at 14mg until End of Treatment (week 26). Throughout the 26 week treatment period, participants in this arm will also take one "sitagliptin placebo" tablet per day.
  Arms: Semaglutide
Drug: Sitagliptin 100mg — participants will take 100mg tablet of Sitagliptin once daily, along with a "semaglutide placebo" pill for the duration of the 26 week treatment period
  Arms: Sitagliptin

SUMMARY:
The effect of once daily dosing of oral Semaglutide versus once daily dosing Sitagliptin on glycemic control, body weight, and safety and tolerability will be compared in Liver Transplant Recipients with poorly-controlled Diabetes Mellitus.

DETAILED DESCRIPTION:
This will be a Phase IV, randomized, parallel, active-controlled, double-blind clinical trial, with one group receiving oral Semaglutide and the other group receiving oral sitagliptin, while continuing any background glucose-lowering medications such as metformin or insulin. Treatment duration will be 26 weeks. Sitagliptin has been chosen as comparator since it is an established oral antidiabetic drug (OAD) within the DPP-4i drug class. There will be a screening period, treatment period, and follow-up period. Furthermore, the investigators will collect biological samples and correlates including serum, plasma, and Intestinal Microbiome samples prior to initiation of study treatment and at the completion of the trial. The investigators will also perform Transient Elastography at these same visits to evaluate change in degree of participant graft steatosis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age ≥18 years at the time of signing informed consent.
* Willing and able to provide informed consent.
* Recipient of liver graft (Liver/Kidney recipients and retransplants allowed)
* Time from transplant surgery ≥ 3 months at time of screening visit with no evidence of active rejection. Liver enzymes must be stable with elevations no greater than 2xULN. However, if patients have elevated liver enzymes beyond 2xULN due to NASH, as confirmed on liver biopsy, they may be included.
* Patient diagnosed with type 2 diabetes or post-transplant diabetes
* Patients transplanted for hepatocellular carcinoma may be included provide their latest surveillance imaging is negative for recurrence
* The use of any immunosuppression regimen (calcineurin inhibitors, mycophenolate mofetil, maintenance prednisone or sirolimus) is acceptable
* HbA1c 7.0-10.5% (53-91 mmol/mol) (both inclusive, not under optimal glycemic control).

Exclusion Criteria:

* Known or suspected hypersensitivity to trial products or related products.
* Previous participation in this trial.
* Active graft dysfunction that requires investigation (at screening).
* Currently receiving steroids (prednisone) for treatment of acute cellular rejection.
* Patients transplanted for multisystem genetic disorders such as amyloidosis or cystic fibrosis.
* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using highly-effective contraceptive methods ().
* Receipt of any investigational medicinal product within 90 days before screening.
* Any disorder or medical condition which, in the investigator's opinion, might jeopardize patient's safety or compliance with the protocol.
* Family or personal history of Multiple Endocrine Neoplasia Type 2 (MEN 2) or Medullary Thyroid Carcinoma (MTC).
* History of pancreatitis (acute or chronic).
* History of major surgical procedures involving the stomach and potentially affecting absorption of trial product (e.g. subtotal and total gastrectomy, sleeve gastrectomy, gastric bypass surgery).
* Any of the following: myocardial infarction (MI), stroke or hospitalization for unstable angina or transient ischemic attack within the past 180 days prior to the day of screening and randomization.
* Classified as being in New York Heart Association (NYHA) Class IV.
* Planned coronary, carotid or peripheral artery revascularization known on the day of screening.
* Renal impairment defined as estimated Glomerular Filtration Rate (eGFR) <30 mL/min/1.73 m2 as per Chronic Kidney Disease Epidemiology Collaboration formula (CKD-EPI).
* Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria in a period of 90 days before the day of screening. An exception is short-term change of insulin treatment for acute illness for a total of ≤ 14 days.
* Known history of proliferative retinopathy or maculopathy requiring acute treatment, unless stable
* History or presence of actively treated malignant neoplasms within the last 5 years (except basal and squamous cell skin cancer, hepatocellular carcinoma, and carcinoma in situ.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c level (%) | Baseline to 26 weeks
  Evaluate the change in glycemic control within and between study groups by measuring HbA1c

SECONDARY OUTCOMES:
Change in body weight (kg) | baseline to 26 weeks
  Evaluate the change in body weight within and between groups
Number of treatment-emergent adverse events | 26 weeks
  safety and tolerability of study drugs.

OTHER OUTCOMES:
Change in aspartate aminotransferase (AST) level | baseline to 26 weeks
  Liver enzyme (AST) level acts as a biomarker of graft injury and will be measured through serum samples during study visits.
Change in alanine aminotransferase (ALT) level | baseline to 26 weeks
  Liver enzyme (ALT) level acts as a biomarker of graft injury and will be measured through serum samples during study visits.

CONTACTS AND LOCATIONS:
Overall Officials: Mamatha Bhat, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No